CLINICAL TRIAL: NCT03076190
Title: Feasibility and Preliminary Efficacy of an Internet-based Pre-surgical Pain Psychology Intervention: A Randomized Controlled Pilot Study of "My Surgical Success"
Brief Title: My Surgical Success: A Randomized Controlled Pilot Study of a Pre-surgical Psychological Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30340
Record Dates: First submitted 2016-12-06; First posted 2017-03-10 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: psychology; pain; surgery; treatment; catastrophizing; cancer
MeSH Terms: conditions — Breast Neoplasms; Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Control Group (Health Education) (No Intervention): Prior to surgery:
  * Demographics survey
  * Baseline surveys
  * Participants receive online information regarding nutrition and exercise that are relevant for people recovering from surgery. Participants are encouraged to incorporate healthy lifestyle choices into their daily routines as they recover from surgery.
  * Follow-up questions about the handouts (detailed above)
  Post-surgery:
  * Daily surveys (detailed above)
  * Follow-up surveys (2, 4, 8, and 12 weeks after surgery)
- My Surgical Success Treatment Group (Experimental): Prior to surgery:
  * Demographics survey
  * Baseline surveys
  * Intervention:
    * 90-minute psychoeducational My Surgical Success video that emphasizes catastrophizing treatment.
    * audio file
    * personalized plan that incorporates the information learned in the video.
  * Follow-up questions about the video (detailed above)
  Post-surgery:
  * Daily surveys (detailed above)
  * Follow-up surveys (2, 4, 8, and 12 weeks after surgery)
  Interventions: Behavioral: Psychoeducational My Surgical Success Video

INTERVENTIONS:
Behavioral: Psychoeducational My Surgical Success Video — The 90-minute video includes instruction by Dr. Beth Darnall, PhD, a pain psychologist at the Stanford Pain Management Center. She teaches the viewer about the relationship between stress, pain, and catastrophizing and provides instruction and skills to reduce catastrophizing, decrease stress, and increase relaxation.
  Arms: My Surgical Success Treatment Group

SUMMARY:
The primary purpose of this study is to determine the feasibility and preliminary efficacy of a remote, Internet-based, pre-surgical psychoeducational intervention delivered to patients scheduled for breast cancer surgery (compared to an active control group that receives health education).

Aim 1: Determine feasibility, satisfaction, and perceived utility of My Surgical Success.

Hypothesis 1: For My Surgical Success, the investigators anticipate 50% engagement in the study (feasibility). Of those who complete My Surgical Success we expect 80% satisfaction ratings, and 80% perceived utility of the information learned.

Aim 2: Determine group differences in within-subject pain catastrophizing scores (baseline - 0 to 48 hours before surgery).

Hypothesis 2: My Surgical Success participants evidence greater reduction in pain catastrophizing (measured with the Pain Catastrophizing Scale; PCS) compared to the HE Control group.

Aim 3: Determine group differences in time to post-surgical pain and opioid cessation.

Hypothesis 3: My Surgical Success participants will evidence quicker time to post-surgical pain and opioid cessation compared to the HE Control Group.

Aim 4: Determine group differences in post-surgical psychological correlates (PROMIS Depression, Anxiety, Function, Pain Interference, Sleep Disturbance, Sleep Related Impairment, Anger, Fatigue, Global, Distress, and Pain Intensity).

Hypothesis 4: My Surgical Success participants will evidence greater post-surgical function and lower pain related interference compared to the HE Control Group.

The goal of this research is to advance our understanding regarding the feasibility and effectiveness of remote psychoeducation interventions and impact on post-surgical outcomes.

DETAILED DESCRIPTION:
Pre-surgical patients are identified by their breast surgeon. The entire study is conducted remotely with no in-person contact with study staff. Study staff call patients and invite them to enroll in the study; informed consent is obtained online.

All participants are asked to provide baseline demographic information, as well as self-reported measures assessing mood, pain, cognitive and emotional responses to pain, catastrophizing, self-efficacy, and medications. All measures are administered via a secure, HIPAA compliant, online system (REDCap).

Participants are then randomized to either the Internet-based pain psychology intervention (My Surgical Success) or to brief online health education (HE Control). Prior to surgery, participants who have been randomized to the HE control group will receive patient handouts online about health and nutrition and are oriented that the information is relevant for improving recovery from surgery. The Internet-based pain psychology intervention emphasizes treatment content that targets pain catastrophizing. My Surgical Success includes a psychoeducational video, a downloadable audio file, and a downloadable PDF Personalized Plan for Success. After viewing the online treatment video, participants randomized to My Surgical Success complete questions regarding participant satisfaction with the video, perceived usefulness of information, and likelihood to use the skills learned. Pain catastrophizing scores are collected from all study participants prior to surgery. All participants are tracked daily post-surgically to assess pain, opioid use, distress, and use of skills learned from treatment; data are captured daily for 30 days, then weekly for 2 weeks, then every 2 weeks for 4 weeks to pain and opioid cessation (or the end of 12 weeks). Psychosocial data are collected post-surgically at weeks 2, 4, 8, and 12.

Post-treatment questions:

Participants in the My Surgical Success group complete the following questions at the end of the video: how understandable the video was, its relevance, usefulness, their satisfaction, how likely they are to use the information, and what they learned from the video.

Participants in HE Control are asked how understandable the health information packet was, its relevance, usefulness, their satisfaction, how likely they are to use the information, and what they learned from the packet.

The pain catastrophizing scale (PCS) is administered following treatment and before surgery to all participants.

Following surgery, all participants fill out online daily measures to assess pain and medication use. Daily measures continue until the participant reports 3 consecutive reports of zero average pain and zero opiate use and has indicated they have recovered from surgery. Until reaching this endpoint, daily measures are collected for 30 days, then bi-weekly for an additional 2 weeks, and then weekly for a period of between 2-6 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Scheduled for breast cancer surgery
* English speaking
* Ability and willingness to complete study procedures including online questionnaires, assessments, and the psychoeducational video

Exclusion Criteria:

* Any conditions causing inability to complete study procedures (e.g. education, cognitive ability, mental status, medical status) or lack of access to internet and phone that would prevent participation in study procedures - at the discretion of the investigator.
* Known pregnancy
* Ongoing legal action related to pain or disability claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth D Darnall, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Darnall BD, Ziadni MS, Krishnamurthy P, Flood P, Heathcote LC, Mackey IG, Taub CJ, Wheeler A. "My Surgical Success": Effect of a Digital Behavioral Pain Medicine Intervention on Time to Opioid Cessation After Breast Cancer Surgery-A Pilot Randomized Controlled Clinical Trial. Pain Med. 2019 Nov 1;20(11):2228-2237. doi: 10.1093/pm/pnz094. PMID 31087093

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants declined to participate; 127 were randomized
Groups:
- My Surgical Success Treatment Group: Prior to surgery:
  * Demographics survey
  * Baseline surveys
  * Intervention:
    * 90-minute psychoeducational My Surgical Success video that emphasizes catastrophizing treatment.
    * audio file
    * personalized plan that incorporates the information learned in the video.
  * Follow-up questions about the video (detailed above)
  Post-surgery:
  * Daily surveys (detailed above)
  * Follow-up surveys (2, 4, 8, and 12 weeks after surgery)
  Psychoeducational My Surgical Success Video: The 90-minute video includes instruction by Dr. Beth Darnall, PhD, a pain psychologist at the Stanford Pain Management Center. She teaches the viewer about the relationship between stress, pain, and catastrophizing and provides instruction and skills to reduce catastrophizing, decrease stress, and increase relaxation.
Period: Overall Study
Arm/Group | Active Control Group (Health Education) | My Surgical Success Treatment Group
Started | 50 | 77
Completed | 32 | 36
Not Completed | 18 | 41
Not completed — Lost to Follow-up | 9 | 34
Not completed — Excluded from Analysis (zero duration ev | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control Group (Health Education) | My Surgical Success Treatment Group | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Categorical [Count of Participants; unit: Participants] — one participant from the control group and 6 participants from the treatment group had missing demographic data Population: Overall number of baseline participants represents the number of participants whose ages we had and are not a reflection of how many participants we collected data on. We had missing demographic data on these participants.
  Participants
    number analyzed (Participants) | 31 | 30 | 61
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 27 | 27 | 54
    >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — One participant from the control group and 6 participants from the treatment group had missing demographic data Population: One participant from the control group and 6 participants from the treatment group had missing demographic data
  years
    number analyzed (Participants) | 31 | 30 | 61
    (all) | 51.16 (11.45) | 51.27 (11.14) | 51.21 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 36 | 68
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 10 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 23 | 20 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 32 | 36 | 68

OUTCOME MEASURES:

1. Primary Outcome: Participant Ratings (0-6) for Satisfaction, Usefulness of the Information Presented, Relevance, Ease of Understanding, and Likelihood to Use Skills Learning
Description: Participants complete a single time point rating for 5 items listed above. Ratings occur on a 0-6 point scale (e.g., 0=completely useless and 6=Very useful). Means and Standard Deviations are reported per the table below.
Time Frame: Immediately post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Control Group: Health Education Active Control Group
- My Surgical Success Treatment Group: My Surgical Success Intervention Group
Arm/Group | Active Control Group | My Surgical Success Treatment Group
Number analyzed (Participants) | 32 | 36
units on a scale
  Easy to Understand | 5.9 (.3) | 5.9 (.2)
  Relevant | 4.7 (1.51) | 5.0 (1.6)
  Useful | 4.67 (1.52) | 5.1 (1.3)
  Satisfaction | 4.67 (1.56) | 5.2 (1.2)
  Likely to Use | 5.03 (1.3) | 5.3 (1.2)

2. Secondary Outcome: Group Difference in Within-subject Pain Catastrophizing
Description: Pain Catastrophizing Scale is a validated 13-item measure assessing levels of pain catastrophizing. Scores range from 0-52, with a higher score indicating higher levels of pain catastrophizing. Data below presents total scores on the scale.
Time Frame: Before surgery to post-surgically
Population: Before Surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control Group | My Surgical Success Treatment Group
Number analyzed (Participants) | 32 | 36
score on a scale | 8.24 (1.19) | 6.62 (1.12)

3. Other Pre Specified Outcome: Group Difference in Time to Opioid Cessation
Description: Postsurgical opioid stop date was self-reported by patients. The opioid stop date was collected through the two-, four-, eight-, and 12-week follow-up surveys with the question "On what date did you stop taking your opioid medication?" The number of postsurgical days using opioids was calculated by subtracting the opioid stop date from the surgery date obtained in the medical chart. Statistical analyses present the data in mean number of days to opioid cessation in each group.
Time Frame: Data on opioid use was collected for the 4 month duration of the study
Measure: Mean (Standard Error); unit: Days to opioid cessation
Arm/Group | Active Control Group | My Surgical Success Treatment Group
Number analyzed (Participants) | 32 | 36
Days to opioid cessation | 21.83 (4.11) | 11.19 (2.21)

4. Other Pre Specified Outcome: Group Difference in Post-surgical PROMIS Physical Function and PROMIS Pain Interference
Description: PROMIS scores for physical function and pain interference will be reported post-surgically. All PROMIS assessments were converted from raw scores to t-scores (Mean= 50, SD=10). Higher scores on PROMIS pain interference signify greater severity of pain interfering with patient's functioning. However, higher scores on Physical function reflects a greater level of physical functioning. The investigators will conduct within subject analyses and will report pre-post treatment changes.
Time Frame: From baseline to post-surgery (up to 4 months duration of the study)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Health Education Control: Health Education active control group
- My Surgical Success: My Surgical Success Intervention Group
Arm/Group | Health Education Control | My Surgical Success
Number analyzed (Participants) | 32 | 36
score on a scale
  Pain Interference | 4.31 (9.65) | 6.77 (9.31)
  Physical Health | 2.56 (6.41) | 0.72 (6.15)

5. Other Pre Specified Outcome: Characterize Responders to My Surgical Success (Demographics and Psychological Correlates)
Description: The investigators will report the baseline psychosocial scores (PROMIS measures) for patients who report high satisfaction with the My Surgical Success treatment. Pain Intensity Scale ranges from 0 (no Pain) to 10 (the worst pain imaginable), with higher scores indicating worse pain. Total scores range from 0-10. Pain Catastrophizing Scale is a 13-item measure assessing levels of pain catastrophizing. Scores range from 0-52, with a higher score indicating higher levels of pain catastrophizing. All PROMIS assessments were converted from raw scores to t-scores (M= 50, SD=10). There are no minimum and maximum values as these are standardized scores. PROMIS Pain Intensity, Pain Interference, Physical Function, Depression, Anxiety, were administered at baseline. Higher scores on PROMIS depression, anxiety, pain interference, and pain intensity signify greater severity of these symptoms. However, higher scores on Physical Function reflects a greater level of physical functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Responders to Treatment: Characterize responders to My Surgical Success (demographics and psychological correlates)
Arm/Group | Responders to Treatment
Number analyzed (Participants) | 36
score on a scale
  Pain Intensity | 1.47 (1.12)
  Pain Catastrophizing | 7.33 (1.3)
  PROMIS physical functioning | 37.52 (5.42)
  PROMIS Pain Interference | 47.49 (1.59)
  PROMIS Anxiety | 54.49 (1.48)
  PROMIS Depression | 47.15 (1.29)

ADVERSE EVENTS:
Time Frame: For the full duration of the study (4 months)
Description: Adverse Event Information was not collected. None of the patients enrolled in the study died during the duration of the study.
Arm/Group | Active Control Group (Health Education) | My Surgical Success Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The sample was underpowered to detect medium effects; Populations with pre-existing pain may better engage in a treatment to address a relevant problem; The study sample was women undergoing surgery for breast cancer, which limits generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-07-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03076190/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03076190/SAP_001.pdf